CLINICAL TRIAL: NCT00875550
Title: A Phase III Randomized, Double-blind, Dose-Controlled, Multicenter Study Evaluating the Safety and Efficacy of Dexmedetomidine in Intubated and Mechanically Ventilated Pediatric Intensive Care Unit Subjects
Brief Title: Study Evaluating Safety and Efficacy of Dexmedetomidine (DEX) in Intubated and Mechanically Ventilated Pediatric Intensive Care Unit (PICU) Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX-08-05
Record Dates: First submitted 2009-03-31; First posted 2009-04-03 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Sedation
Keywords: Intubated and mechanically ventilated PICU subjects
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine Low Dose (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Fentanyl; Drug: Morphine
- Dexmedetomidine High dose (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Fentanyl; Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine — Study drug titrated up or down to maintain target UMSS range.
Drug: Midazolam — Rescue medication for sedation according to UMSS scores
Drug: Fentanyl — Rescue medication for pain based on UMSS scores
Drug: Morphine — Rescue medication for pain based on UMSS scores.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of dexmedetomidine (DEX) in intubated and mechanically ventilated pediatric intensive care unit (PICU) subjects. The key study objectives are:

* To characterize the loading and maintenance dosing of DEX by age group and overall medical condition of pediatric subjects
* To evaluate the safety and efficacy of loading and maintenance infusions for sedation in initially intubated and mechanically ventilated PICU subjects
* To explore the exposure-response relationship between dose of DEX and clinical measures of sedation and safety

DETAILED DESCRIPTION:
An estimated 175 subjects will be enrolled at approximately 40 investigative sites. Subjects will be divided into two treatment groups to receive either high dose or low dose Dexmedetomidine (DEX). The loading and maintenance doses in both groups will be stratified according to the presence or absence of cardiopulmonary bypass. The level of sedation will be assessed using the University of Michigan Sedation Scale (UMSS). Score 0 (awake/alert); Score 1 (sleepy/responds appropriately); Score 2 (somnolent/arouses to light stimuli); Score 3 (deep sleep/arouses to deeper); Score 4 (unarousable to stimuli).

Based on these scores and clinical judgment, additional sedation with intravenous midazolam will be administered according to the label. The UMSS scores must be documented before the administration of every midazolam (MDZ) dose and within five minutes after each dose of MDZ. Fentanyl or morphine may be administered to treat pain. Subjects may be extubated after beginning of study drug but are not required to be as part of the study.

The efficacy and safety parameters that will be monitored include sedation levels, heart rate, blood pressure and ventilation indicators. Once subjects have met site-specified respiratory criteria, they will undergo tracheal extubation. The dexmedetomidine infusion may be continued during and after extubation if further sedation is required post-extubation. The continuous infusion of dexmedetomidine must be administered for a minimum of 6 hours and a maximum of 24 hours. Sedation levels, heart rate, blood pressure, respiratory rate, ventilator settings, SpO2 and if available transcutaneous carbon dioxide (TcCO2) and/or arterial blood gases (ABG) will be monitored and recorded in the peri-extubation period.

ELIGIBILITY:
Inclusion Criteria:

1. Initially intubated and mechanically ventilated pediatric subjects (≥1 month [birth age corrected for prematurity] to <17 years of age) in an intensive care setting. The means by which the subject is intubated may include nasotracheal, endotracheal or via tracheotomy. The subject must be mechanically ventilated prior to and during the commencement of study drug.
2. Anticipated to require a minimum of 6 hours of continuous intravenous sedation.
3. American Society of Anesthesiologists (ASA) classification of 1, 2, 3 or 4.
4. A UMSS score of 1, 2, 3 or 4 at the start of infusion of study drug.
5. A dose has been established for this subject's age based upon the diagnosis procedures.

   Status post cardiopulmonary bypass (s/p CPB):
   * Low dose group: Loading dose: 0.2 mcg/kg Maintenance dose titration range (0.025-0.5 mcg/kg/hr)
   * High dose group: Loading dose: 0.5 mcg/kg Maintenance dose titration range (0.1-0.7 mcg/kg/hr)

   All other diagnoses:
   * Low dose group: Loading dose: 0.3 mcg/kg Maintenance dose titration range (0.05- 0.5mcg/kg/hr)
   * High dose group: Loading dose: 0.6 mcg/kg Maintenance dose titration range (0.2 - 1.4 mcg/kg/hr)
6. If female, subject is non-lactating and is either:

   1. Not of childbearing potential, defined as pre-menarche, or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
   2. Of childbearing potential but is not pregnant at time of baseline.
7. Subject's parent(s) or legal guardian(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board. Assent will be obtained where age-appropriate and according to state regulations.

Exclusion Criteria:

1. Pediatric subjects with neurological conditions that prohibit an evaluation of sedation in the opinion of the investigator (e.g. increased intracranial pressure or extensive brain surgery).
2. The infusion pump minimal capacity cannot accommodate the lowest possible maintenance infusion rate of study drug based on subject's weight.
3. Subjects with second degree or third degree heart block unless subject has a pacemaker or pacing wires.
4. Hypotension that persist beyond a 15 min of re-assessments prior to starting study drug:

   * Age 1 month to ≤6 months old: systolic blood pressure (SBP) <60 (millimeters of mercury) mmHg
   * Age >6 months to <2 yrs old: SBP <70 mmHg
   * Age >2 to <12 yrs old: SBP <80 mmHg
   * Age >12 to <17 yrs old: SBP <90 mmHg
5. Pre-existing bradycardia that persists beyond a 15 min period of re-assessment prior to starting study drugs:

   * Age 1 month to <2 months old: HR <90 beats per min (bpm)
   * Age ≥2 months to <12 months old: HR <80 bpm
   * Age ≥12 months to <2 yrs old: HR <70 bpm
   * Age ≥ 2 to <12 yrs old: HR <60 bpm
   * Age ≥ 12 to <17 yrs old: HR <50 bpm
6. Serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT): 1 month -12 months: >165 U/L; >12 months to <17 years: ≥100 U/L.

   Note: Subjects may be rescreened up to 6 hrs prior to study drug infusion (not including subjects undergoing cardiac surgery with CPB).
7. Subjects who have a known allergy to dexmedetomidine, MDZ, morphine or fentanyl.
8. Requirement for medications other than DEX, midazolam, morphine or fentanyl for sedation and pain control.
9. Subjects with immobility form neuromuscular disease, paralysis from administration of neuromuscular blocking agents, spinal cord injury above T5, or subjects with muscle weakness form congenital or systemic medical illness etiologies. Note: subjects who received NMB agents intraoperatively must be, in the Investigator's opinion, free of residual neuromuscular blockade prior to dosing with study drug.
10. Subjects who have received another investigational drug or device within the past 30 days.
11. Subjects who have received DEX in a previous investigational trial within the previous 12 weeks.
12. Subjects who, in the opinion of the investigator, have any other condition where the risks of DEX would be expected to outweigh its benefits (e.g. cardiogenic shock on >2 vasopressors).
13. Subjects who will require alpha-2 agonists/antagonists listed below within 48 hrs prior to baseline.

Alpha-2 Agonists: Xylazine*, Clonidine (Catapres, Dixarit), Guanfacine (Tenex), Guanabenz (Wytensin), Mivazerol, Guanadrel (Hylorel), Guanethidine (Ismelin) and Methyldopa (Aldomet). * Xylazine is a veterinary product, but has abuse potentIal in humans.

Alpha-2 Antagonists: Corynanthine, Phenoxybenzamine (Dibenzyline), Phentolamine (Regitine, Rogitine), Tolazoline (Priscoline), Yohimbine, Rauwolscine, Idazoxan, Reserpine (Serpasil) and Mirtazapine (Remeron, Remeron Soltab).

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bilkovski, MD, Study Director — Medical Director, Hospira
Locations (37):
- United States (33):
  - Maricopa Medical Center, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Pediatric Dept., Div. of Critical Care - PICU, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Pediatric Critical Care, Los Angeles, California
  - Dept. of Anesthesia, SUMC, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Joe Dimaggio Children's Hospital/Memorial Regional Hospital, Pediatric Intensive Care Unit, Hollywood, Florida
  - Critical Care, Jacksonville, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Orlando, Florida
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Children's Hospital, Park Ridge, Illinois
  - Kosair Charities Pediatric Clinical Research Unit, University of Louisville, Louisville, Kentucky
  - The John Hopkins Medical Institutions, Anesthesia and Critical Care Medicine, Baltimore, Maryland
  - F3900 C.S. Mott Hospital SPC 5211 Dept. of Anaesthesiology, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Gilette Children's Speciality Healthcare, Saint Paul, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Department of Anesthesiology, Durham, North Carolina
  - Akron Children's Hospital Medical Center, Akron, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Northwest Pediatric Critical Care, P.C. Legacy Emanuel Children's Hospital, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Virginia, Division of Pediatric Critical Care, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Madison, Wisconsin
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Pediatric Intensive Care Unit, CHU Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine Low Dose: Dexmedetomidine: Loading dose 0.2 mcg/kg or 0.3 mcg/kg, Maintenance dose titration range (0.025-0.5 mcg/kg/hr) or (0.05-0.5 mcg/kg/hr)
  Midazolam: Rescue medication for sedation according to UMSS scores
  Fentanyl: Rescue medication for pain based on UMSS scores
  Morphine: Rescue medication for pain based on UMSS scores.
- Dexmedetomidine High Dose: Dexmedetomidine: Loading dose 0.5 mcg/kg or 0.6 mcg/kg, Maintenance dose titration range (0.1-0.7 mcg/kg/hr) or (0.2-1.4 mcg/kg/hr)
  Midazolam: Rescue medication for sedation according to UMSS scores
  Fentanyl: Rescue medication for pain based on UMSS scores
  Morphine: Rescue medication for pain based on UMSS scores.
Period: Overall Study
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Started | 89 | 86
Completed | 77 | 76
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose | Total
Number analyzed (Participants) | 89 | 86 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.35 (3.437) | 2.85 (4.172) | 2.60 (3.814)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89 | 86 | 175
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Number; unit: participants]
  >= 1 month to < 24 months | 63 | 60 | 123
  >=24 months to < 17 years old | 26 | 26 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 53 | 48 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 14 | 28
  White | 64 | 62 | 126
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 7 | 3 | 10
American Society of Anaesthesiologists (ASA) classification [Number; unit: participants]
  P1 - Normal healthy patient (PT) | 3 | 5 | 8
  P2 - PT w/ mild systemic disease | 28 | 16 | 44
  P3 - PT w/ severe systemic disease) | 50 | 53 | 103
  P4 - PT w/ constant threat to life) | 8 | 12 | 20
  P5 - Moribund patient | 0 | 0 | 0
  P6 - A declared brain-dead patient | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That do Not Require Rescue Midazolam (MDZ) for Sedation Based on Achieving and Maintaining a Target University of Michigan Sedation Scale (UMSS) Score of 1 to 3 While Intubated.
Description: Clinical Score Level of Sedation 0 Awake/Alert
  1. Minimally Sedated: Tired/sleepy, appropriate response to verbal conversation and/or sounds.
  2. Moderately Sedated: Somnolent/sleeping, easily aroused with light tactile stimulation.
  3. Deeply sedated: Deep sleep, arousable only with significant physical stimulation.
  4. Unarousable
Time Frame: 6 to 24 hours
Population: Efficacy Evaluable Population: All subjects randomized to study medication and who received randomized DEX for at least 6 hours
Measure: Number; unit: Percentage of subjects
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
Percentage of subjects | 44.6 | 54.3

2. Secondary Outcome: Absolute Time on Study Drug That the Subject is in a UMSS Range of 1 to 3 While Intubated
Time Frame: 6 to 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
Hours | 17.2 [5 to 24] | 17.3 [2 to 24]

3. Secondary Outcome: Absolute Time on Study Drug That the Subject is Out of the Target Sedation Range (UMSS <1 or >3) While Intubated
Time Frame: 6 to 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
hours | 1.0 [0 to 10] | 0.7 [0 to 14]

4. Secondary Outcome: Total Amount of Rescue Medication Required for Sedation and Analgesia While Intubated
Time Frame: 6 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
Milligram
  Midazolam | 2.221 (4.6089) | 1.241 (2.3052)
  Fentanyl | 45.225 (83.7743) | 44.367 (112.13)
  Morphine | 1.446 (3.2978) | 1.141 (2.4209)

5. Secondary Outcome: Time to First Dose of Rescue Medication for Sedation and Analgesia
Time Frame: 6 to 24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
Hours | 1.6 [0.933 to 3.383] | 2.0 [1.067 to 3.750]

6. Secondary Outcome: Time to Successful Extubation
Time Frame: 6 to 24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Number analyzed (Participants) | 83 | 81
Hours | 23.8 [18.550 to NA] — Computation for the 95% confidence interval (CI) from the Kaplan-Meier analysis requires adequate number of events to be estimable. There were not enough events to fully characterize the complete CI, only point estimate and the 95% lower CI estimate. | 20.5 [17.133 to 23.333]

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine Low Dose | Dexmedetomidine High Dose
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/86
Other Adverse Events (participants affected / at risk) | 48/89 | 43/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Low Dose (N=89) | Dexmedetomidine High Dose (N=86)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine Low Dose (N=89) | Dexmedetomidine High Dose (N=86)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 3
Extrasystoles (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4
Chest pain (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 2 | 0
General symptom (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 7 | 5
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Device electrical finding (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Base excess decreased (Investigations) | 1 | 0
Blood albumin abnormal (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood cortisol increased (Investigations) | 0 | 1
Blood culture positive (Investigations) | 1 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Blood magnesium abnormal (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 1
Blood pH decreased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 2 | 2
Blood potassium abnormal (Investigations) | 1 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 1
Carbon dioxide decreased (Investigations) | 1 | 0
Central venous pressure decreased (Investigations) | 0 | 1
Culture positive (Investigations) | 0 | 1
Culture urine positive (Investigations) | 0 | 1
Electrocardiogram (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 2
Haematocrit decreased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Heart rate decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 2 | 0
Oxygen saturation decreased (Investigations) | 1 | 3
PCO2 increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Platelet count increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Respiratory rate decreased (Investigations) | 2 | 0
Sputum culture positive (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0
Crying (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 0
Hypotension (Vascular disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No